CLINICAL TRIAL: NCT00448357
Title: Allogeneic Hematopoietic Cell Transplantation for Patients With Hematologic Disorders Who Are Undergoing Dose-Adjusted Treatment With A Maximally Intensive Busulfex-Based Therapeutic Regimen
Brief Title: Allogeneic Hematopoietic Cell Transplantation for Patients With Busulfex-based Regimen
Acronym: LCCC0510
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0510; P30CA016086 (NIH); NCT00618306 (obsolete NCT alias)
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-06

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage II multiple myeloma; stage III multiple myeloma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; Waldenstrom macroglobulinemia; accelerated phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic neutrophilic leukemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); primary myelofibrosis; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; secondary myelodysplastic syndromes; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; adult acute lymphoblastic leukemia in remission; polycythemia vera; essential thrombocythemia; splenic marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I multiple myeloma; recurrent adult grade III lymphomatoid granulomatosis; adult nasal type extranodal natural killer (NK)/T-cell lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Congenital Abnormalities; Primary Myelofibrosis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Prolymphocytic; Leukemia, Myeloid, Acute; Polycythemia Vera; Thrombocythemia, Essential; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Lymphoma, Extranodal NK-T-Cell | interventions — Antilymphocyte Serum; Busulfan; fludarabine phosphate; Tacrolimus; Peripheral Blood Stem Cell Transplantation; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GVHD prophylaxis (Experimental): Subjects with matched-related donors (MRDs) were treated with tacrolimus and methotrexate with or without alemtuzumab for graft vs host disease prophylaxis Subjects also receive busulfan and fludarabine .
  Matched unrelated donor (MUD) or mismatched related donor (MMRD) subjects receive GVHD prophylaxis with rabbit anti-thymocyte globulin (ATG) + Methotrexate Subjects also receive busulfan, fludarabine, and tacrolimus.
  Interventions: Biological: rabbit anti-thymocyte globulin (ATG); Biological: therapeutic allogeneic lymphocytes; Drug: busulfan; Drug: fludarabine phosphate; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: methotrexate

INTERVENTIONS:
Biological: rabbit anti-thymocyte globulin (ATG) — .5 mg/kg on day -3 and 2.5 mg/kg on day -2
Biological: therapeutic allogeneic lymphocytes — minimum total cluster of differentiation (CD34+) cells of 3 x 10^6 cells/kg and a maximum of 8 x 10^6 cells/kg will be infused on day 0
Drug: busulfan — PK-targeted continuous IV infusion over 90 hours on Days -7 to -4.
Drug: fludarabine phosphate — 30 mg/m^2/day x 5 days intravenous piggyback (IVPB) over 30 minutes on Days -7 through -3
Drug: tacrolimus — The suggested starting dose is 0.03 mg/kg po bid starting on day -1
Procedure: allogeneic hematopoietic stem cell transplantation — A minimum total CD34+ cell dose of 3 x 10^6 cells/kg and maximum of 8 x 10^6 cells/kg will be infused on day 0
Procedure: peripheral blood stem cell transplantation — minimum total CD34+ cell dose of 3 x 10^6 cells/kg and a maximum of 8 x 10^6 cells/kg will be infused on day 0
Drug: methotrexate — 5 mg/m^2 on days +1, +3 and +6

SUMMARY:
RATIONALE: Giving chemotherapy, such as fludarabine and busulfan, before a donor peripheral stem cell transplant helps stop the growth of cancer or abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving a monoclonal antibody, alemtuzumab, before the transplant and tacrolimus after the transplant may stop this from happening.

PURPOSE: The phase I portion of this trial identified the maximum tolerated dose of busulfan after treating 40 patients on a dose-escalation scheme. We are now treating an additional 26 patients on the phase II portion of the trial at a Pharmacokinetic (PK)-directed dose of total area under curve (AUC) 6912 micrometer (uM)-min/24 hours. We transitioned to the Phase II portion of the study in October 2009.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Phase I Objective: To identify the maximum tolerated dose of continuous infusion IV busulfan based on blood levels derived from a test dose in conjunction with fludarabine, ATG and methotrexate plus tacrolimus for GVHD prophylaxis
* Phase II Objective: To determine the one-year disease-free survival (DFS) rate at the maximum tolerated dose identified during Phase I of the trial (target AUC 6912)

Secondary

* Determine the overall and disease-free survival of patients treated with this regimen.
* Determine the dose-limiting toxicities of this regimen in these patients.
* Determine the capacity of test dosing of busulfan that would result in the desired area under the curve concentration exposure of patients receiving a full-dose busulfan regimen.
* Determine the incidence of graft-vs-host disease and DNA chimerism between 1 month and 2 years post-transplantation in these patients.
* Compare the overall survival (OS) and disease-free survival (DFS) rates for patients treated with Campath vs. patients treated with ATG/Methotrexate for GVHD control

OUTLINE: This is a non-randomized, open-label, parallel group study of busulfan. Patients are stratified according to donor relationship - matched related donor (MRD) vs matched unrelated donor (MUD).

* Conditioning regimen: Patients receive fludarabine phosphate IV over 30 minutes on days -7 to -3 and busulfan IV over 2 hours once within days -15 to -10 and then IV continuously over 90 hours on days -7 to -4. Patients with a MRD also receive Methotrexate (MTX) on Days +1, +3, and +6. Patients with a MUD receive ATG on Days -3 and -2 and MTX on Days +1, +3 and +6.

Phase I portion only: Cohorts of 3-6 patients receive escalating doses of busulfan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Allogeneic peripheral blood stem cell transplantation: Patients undergo allogeneic peripheral blood stem cell transplantation on day 0. Patients then receive sargramostim (GM-CSF) subcutaneously beginning on day 5 and continuing until blood counts recover.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive oral tacrolimus twice daily on days -1 to 180 or days -1 to 240.
* Donor lymphocyte infusion (DLI): Patients who do not achieve CR, do not have GVHD, and have been off immunosuppressants for at least 30 days may receive up to 3 DLIs, at least 8 weeks apart, after completion of tacrolimus.

After the completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
INCLUSION CRITERIA

Histologically confirmed diagnosis of any of the following:

Chronic lymphocytic leukemia or prolymphocytic leukemia Chemotherapy-refractory or advanced disease after ≥ 3 prior treatments Chronic myelogenous leukemia Diagnosis based on t(9;22) or related t(9;12) cytogenetic abnormalities AND characterized by elevated white blood counts (WBC) in peripheral blood or marrow Patients with progressive disease on imatinib mesylate or other protein tyrosine kinase inhibitors; less than a major cytogenetic or fluorescent in situ hybridization (FISH) complete response (CR) after a minimum of 6 months of targeted therapy; or less than a complete FISH or cytogenetic response after 12 months of targeted therapy are eligible Patients with other cytogenetic abnormalities, such as t(9;12), that are associated with an aggressive clinical course are eligible Non-Hodgkin's lymphoma (NHL) or Hodgkin's lymphoma Any World Health Organization (WHO) classification histologic subtype allowed Must have advanced disease as defined by relapse after initial CR or failure to achieve CR OR deemed to have less than a 30% likelihood of durable response with an autologous stem cell transplant Refractory low-grade NHL histologies or any intermediate or aggressive large cell or mantle cell lymphoma allowed Acute myeloid leukemia (AML) High-risk disease in first CR (CR1) OR evidence of any recurrent disease beyond CR1 High-risk individuals are those requiring more than 1 course of induction therapy to achieve remission; those with extra-medullary disease at presentation; or those with high-risk cytogenetic abnormalities (abnormalities of chromosomes 5, 7, 2, trisomy 8, or 3) or > 2 cytogenetic abnormalities

* Multiple myeloma
* Myelodysplastic syndromes (MDS) Must have MDS defined by WHO criteria with > 5% blasts or high-risk cytogenetic abnormalities (abnormalities of chromosomes 5, 7, 2, trisomy 8, or 3)
* Acute lymphoblastic leukemia (ALL) High-risk disease in CR1 OR beyond CR1 High-risk disease includes the following: t(9;22) or t(4;11); WBC > 30,000/mm³ at presentation; non-T-cell phenotype; or more than 30 years of age
* Myelofibrosis/agnogenic myeloid metaplasia

  * Patients must be transfusion dependant or have evidence of evolving AML as evidenced by an excess of blasts or a state of marrow failure/fibrosis
  * Myeloproliferative disorders with advanced disease (e.g., progressive or spent phase polycythemia vera, myelofibrosis, or essential thrombocythemia)

    * Any of the following categories of donors are acceptable*:
* Human Leucocyte Antigen (HLA)-identical or 1 antigen-mismatched sibling (5/6, 6/6, or 8/10) donor

  * Minimal serologic typing required for class I (A, B); molecular typing required for class II (DRB1)
* 8/10 matched unrelated donor (MUD)

  * Molecular analysis at HLA-A, -B, -C, -DRB1 and -DQB1 (8/10 match) by high resolution typing is required
* 5/6 MUD

  * Molecular analysis at HLA-A, -B, and -DRB1 required Note: *No syngeneic donors

PATIENT CHARACTERISTICS:

* Performance status 0-2
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2 times ULN
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Diffusing capacity of the lungs for carbon monoxide (DLCO) > 60% with no symptomatic pulmonary disease
* Left ventricular ejection fraction (LVEF) ≥ 50% by multigated acquisition (MUGA) scan

EXCLUSION CRITERIA Uncontrolled or severe cardiovascular disease, pulmonary disease, or infection that, in the opinion of the treating physician, would make this study unreasonably hazardous to the patient Other serious illness that would limit survival to < 2 years Psychiatric condition that would preclude study compliance Uncontrolled diabetes mellitus or active serious infection Active second malignancy except for nonmelanomatous skin cancer Known hypersensitivity to E. coli-derived products HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy, radiotherapy, or surgery

  * Cranial radiotherapy or intrathecal therapy as prophylaxis against central nervous system (CNS) recurrence within the past 4 weeks allowed (in high-risk patients)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2005-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Shea, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shea TC, Walko C, Chung Y, Ivanova A, Sheets J, Rao K, Gabriel D, Comeau T, Wood W, Coghill J, Armistead P, Sarantopoulos S, Serody J. Phase I/II Trial of Dose-Escalated Busulfan Delivered by Prolonged Continuous Infusion in Allogeneic Transplant Patients. Biol Blood Marrow Transplant. 2015 Dec;21(12):2129-2135. doi: 10.1016/j.bbmt.2015.07.016. Epub 2015 Jul 22. PMID 26210442
- See also: University of North Carolina Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with advanced, refractory, or high-risk hematologic cancers who were deemed suitable for myeloablative conditioning were recruited from one institution.
Pre-assignment Details: A total of 55 subjects were consented, but one subject was not enrolled due to disease progression or death prior to protocol therapy.
Groups:
- Experimental: GVHD Prophylaxis: Experimental: GVHD prophylaxis
  Subjects with matched-related donors (MRDs) were treated with tacrolimus and methotrexate with or without alemtuzumab for graft vs host disease prophylaxis Subjects also receive busulfan and fludarabine .
  Matched unrelated donor (MUD) or mismatched related donor (MMRD) subjects receive GVHD prophylaxis with rabbit anti-thymocyte globulin (ATG) + Methotrexate Subjects also receive busulfan, fludarabine, and tacrolimus.
Period: Overall Study
Arm/Group | Experimental: GVHD Prophylaxis
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: GVHD Prophylaxis
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 50 [27 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 48
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 54
Donor-recipient sex [Count of Participants; unit: Participants]
  Male-Female | 6
  Female-Male | 12
  Male-Male | 22
  Female-Female | 14
Host cytomegalovirus (CMV) status [Count of Participants; unit: Participants]
  Negative | 18
  Positive | 36
Disease histology [Count of Participants; unit: Participants]
  Myelogenous leukemia | 26
  Myelodysplasia | 8
  Chronic myelogenous leukemia | 1
  Acute lymphoblastic leukemia | 7
  Non-Hodgkin Lymphoma | 5
  Hodgkin lymphoma | 2
  Myelofibrosis | 1
  Chronic lymphoblastic leukemia | 1
  Chronic myelomonocytic leukemia | 1
  Plastic cell leukemia | 2
Type of transplant [Count of Participants; unit: Participants]
  Matched unrelated donor (MUD) | 34
  Matched unrelated donor (MRD) | 20
Disease risk [Count of Participants; unit: Participants]
  Low | 16
  Intermediate | 20
  High | 18

OUTCOME MEASURES:

1. Primary Outcome: Three-year Relapse-free Survival (RFS) Rate at the Maximum Tolerated Dose Identified During Phase I of the Trial (Target AUC 6912)
Description: Relapse is defined as new or increased sites of disease or positive one marrow after a complete response (CR). The RFS was calculated as the percentage of patients who were alive and without relapse at 3 years
Time Frame: Three years post-transplant
Population: Because AUC levels varied between the groups and the goal was to identify an actual achieved AUC-based dose, additional outcome analyses were undertaken by dividing patients into thirds according to the actual AUCs delivered rather than the original planned AUCs.
Measure: Number; unit: percentage of participants
Groups:
- Low Busulfan AUC Tertile: Participants with the lowest tertile of measured busulfan Area under the curve (AUC); with a mean value of 5078 (full range 3933-5615) microM/min
- Intermediate Busulfan AUC Tertile: Participants with the lowest tertile of measured busulfan Area under the curve (AUC); with a mean value of 6372 (full range 5639-6965) microM/min
- High Busulfan AUC Tertile: Participants with the lowest tertile of measured busulfan Area under the curve (AUC); with a mean value of 7605 (full range 7054-8863) microM/min
Arm/Group | Low Busulfan AUC Tertile | Intermediate Busulfan AUC Tertile | High Busulfan AUC Tertile
Number analyzed (Participants) | 18 | 18 | 18
percentage of participants | 22 | 39 | 43

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Dose limiting toxicity will be defined as any irreversible grade 3 or any grade 4 non-hematologic toxicity that is related to busulfan infusion and not graft vs host disease or late infection after recovery from the initial period of myelosuppression. The maximum tolerated dose (MTD) is defined as the dose with probability of dose limiting toxicity (DLT) of 0.25. The dose of continuous infusion IV busulfan based on blood levels derived from a test dose in conjunction with fludarabine and alemtuzumab plus tacrolimus for GVHD prophylaxis.
Time Frame: first 6 weeks or 42 days following stem cell infusion
Measure: Number; unit: DLTs
Groups:
- Dose Level 1: Target AUC/24 hrs of 4800 micrometer (uM)-min +/-15%
- Dose Level 2: Target AUC/24 hrs of 5760 uM-min +/- 15%
- Dose Level 3: Target AUC/24 hrs of 6912 uM-min +/- 15%
- Dose Level 4: Target AUC/24 hrs of 7603 uM-min+/- 15%
- Dose Level 5: Target AUC/24 hrs of 8363 uM-min+/- 15%
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 14 | 7 | 24 | 7 | 2
DLTs | 1 | 1 | 1 | 2 | 2

3. Secondary Outcome: Capacity of Test Dosing of Busulfan That Would Result in the Desired Area Under the Curve Concentration Exposure of Patients Receiving a Full-dose Busulfan Regimen
Description: Test doses of busulfan were administered and plasma levels were measured to determine a targeted AUC dosing estimate. The capacity is reported as the precision with which these test dose goals predicted the actual 90-hour mean AUC levels.Dose targeting precision was estimated by root mean squared error.
Time Frame: Day -15 to Day -11
Measure: Number; unit: percentage of error
Groups:
- Dose Level 1: Target AUC/24 hrs of 4800 uM-min +/-15%
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 14 | 7 | 24 | 7 | 2
percentage of error | 11.7 | 4.9 | 10.2 | 11.1 | 15.9

4. Secondary Outcome: Incidence of Graft vs Host Disease in Patients Between One Month and Two Years Post Transplant
Description: GVHD can be mild, moderate or severe depending on the differences in tissue type between patient and donor. GVHD can be acute or chronic. Its symptoms can include:
  * Rashes, which include burning and redness, that erupt on the palms or soles and may spread to the trunk and eventually to the entire body
  * Blistering, causing the exposed skin surface to flake off in severe cases
  * Nausea, vomiting, abdominal cramps, diarrhea and loss of appetite, which can indicate that the gastrointestinal (digestive) tract is affected
  * Jaundice, or a yellowing of the skin, which can indicate liver damage
  * Excessive dryness of the mouth and throat, leading to ulcers
  * Dryness of the lungs, vagina and other surfaces
Time Frame: 100 days post transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Busulfan AUC Tertile | Intermediate Busulfan AUC Tertile | High Busulfan AUC Tertile
Number analyzed (Participants) | 18 | 18 | 18
Participants
  Acute GVHD grade >=II | 7 | 10 | 11
  Acute GVHD grades III and IV | 2 | 4 | 3
  Chronic GVHD; intermediate/severe | 4 | 6 | 2

5. Secondary Outcome: Incidence of DNA Chimerism in Patients Between One Month Post Transplant
Description: Deoxyribonucleic acid (DNA) chimerism is a measure identifying the genetic profiles of the transplant recipient and of the donor and then evaluating the extent of mixture in the recipient's blood, bone marrow, or other tissue.
Time Frame: 30 days post transplant
Population: Because there were no differences in chimerism results as a function of either the immunosuppression used or busulfan dose received, the results are being reported only for the total population.
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: GVHD Prophylaxis: Matched related donor (MRD) subjects receive Graft Vs Host Disease (GVHD )prophylaxis with Methotrexate alone Subjects also receive busulfan, fludarabine, and tacrolimus and may receive Alemtuzumab.
  Matched unrelated donor (MUD) or mismatched related donor (MMRD) subjects receive GVHD prophylaxis with rabbit anti-thymocyte globulin (ATG) + Methotrexate Subjects also receive busulfan, fludarabine, and tacrolimus.
Arm/Group | Experimental: GVHD Prophylaxis
Number analyzed (Participants) | 54
Participants
  Whole blood chimerism-Any | 49
  Whole blood chimerism->=95% donor | 47
  T Cell chimerism-Any | 46
  T Cell chimerism>=95% donor | 30

6. Secondary Outcome: Overall Survival
Description: Percentage of participants alive at 3 years post transplant
Time Frame: Three years post-transplant
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Low Busulfan AUC Tertile (5078): Participants with the lowest tertile of measured busulfan Area under the curve (AUC); with a mean value of 5078 (full range 3933-5615) microM/min
- Intermediate Busulfan AUC Tertile (6372): Participants with the lowest tertile of measured busulfan Area under the curve (AUC); with a mean value of 6372 (full range 5639-6965) microM/min
- High Busulfan AUC Tertile (7605): Participants with the lowest tertile of measured busulfan Area under the curve (AUC); with a mean value of 7605 (full range 7054-8863) microM/min
Arm/Group | Low Busulfan AUC Tertile (5078) | Intermediate Busulfan AUC Tertile (6372) | High Busulfan AUC Tertile (7605)
Number analyzed (Participants) | 18 | 18 | 18
percentage of participants | 28 | 39 | 55

ADVERSE EVENTS:
Time Frame: Mortality was assessed at one year
Description: Additional toxicities were not captured as this was a high-dose transplant study and grades 1, 2 and 3 AEs were generally expected and no unexpected toxicities were seen beyond those reported as SAEs
Arm/Group | Experimental: GVHD Prophylaxis
All-Cause Mortality (participants affected / at risk) | 15/54
Serious Adverse Events (participants affected / at risk) | 26/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: GVHD Prophylaxis (N=54)
BK cystitis (Infections and infestations) | 1
Liver Failiure (Hepatobiliary disorders) | 1
Sepsis (Infections and infestations) | 4
Gr 4 GVHD (Gastrointestinal disorders) | 1
Gr 4 mucositis (Gastrointestinal disorders) | 5
Veno-occlusive disease (Hepatobiliary disorders) | 3
Aspergillus pneumonia (Infections and infestations) | 2
CMV pneumonitis (Infections and infestations) | 1
Graft Failure (Blood and lymphatic system disorders) | 1
Diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
anemia (Blood and lymphatic system disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 4
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
renal Failure (Renal and urinary disorders) | 2
left neck hematoma (Vascular disorders) | 1
Glucose Intolerance (Endocrine disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: GVHD Prophylaxis (N=54)
grade 3 or 4 hematologic toxicities (expected) (Blood and lymphatic system disorders) | 54 — Additional toxicities were not captured as this was a high-dose transplant study and grades 1, 2 and 3 adverse events (AEs) were generally expected and no unexpected toxicities were seen beyond those reported as Serious Adverse Events (SAEs)
Alopecia (Skin and subcutaneous tissue disorders) | 54
grade 3 GI toxicity (Gastrointestinal disorders) | 21 — nausea or diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes